CLINICAL TRIAL: NCT00668707
Title: Adjuvant Melatonin for Prevention of Lung Cancer Recurrence and Mortality: A Randomized Placebo Controlled Clinical Trial
Brief Title: Adjuvant Melatonin for Prevention of Lung Cancer Recurrence and Mortality
Acronym: AMPLCaRe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: The Ottawa Hospital (Other); Lotte & John Hecht Memorial Foundation (Other); Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007077-01H
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: melatonin; natural health product (NHP); lung cancer; complementary and alternative medicine (CAM); randomized clinical trial
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): To receive 20 mg of melatonin nightly for 1 year post-surgery
  Interventions: Dietary Supplement: melatonin
- Placebo (Placebo Comparator): To receive 20 mg placebo nightly for 1 year post-surgery
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: melatonin — 20 mgs ingested nightly
  Arms: Melatonin
Dietary Supplement: placebo — similar to experimental in all ways except for lack of active ingredient
  Arms: Placebo

SUMMARY:
There is evidence to support the use of melatonin, a natural health product, as an additional treatment aid for cancer patients. This study is designed to see if the daily ingestion of 20 milligrams of melatonin for one year can lower the incidence of developing lung cancer recurrence and/or death. Only patients with a diagnosis of non small cell lung cancer who are eligible for surgical resection can participate in the trial. The study will also be assessing for changes in quality of life, pain, fatigue, anxiety, sleep, and depression amongst the participants.

DETAILED DESCRIPTION:
The trial employs a two-armed parallel placebo controlled trial design whereby patients with a diagnosis of non small cell lung cancer are randomized to receive either 20 mg of melatonin nightly or an identically matched placebo. All patients will be followed for two years with primary outcomes assessed at a two year time point and secondary outcomes evaluated throughout the course of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non small cell lung cancer
* Eligible for surgical resection
* Willingness to adhere to randomized treatment
* Availability for follow-up schedule of visits

Exclusion Criteria:

* Taking exogenous melatonin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2007-09; Primary Completion 2017-03-09 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dugald MR Seely, ND, MSc, Principal Investigator — The Canadian College of Naturopathic Medicine; Andrew JE Seely, MD, Principal Investigator — The Ottawa Hospital
Locations (8):
- Canada (8):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Fraser Health, Surrey, British Columbia
  - QEII Health Sciences Centre/Capital Health, Halifax, Nova Scotia
  - St. Joseph's/ McMaster University, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec

REFERENCES:
- [Background] Mills E, Wu P, Seely D, Guyatt G. Melatonin in the treatment of cancer: a systematic review of randomized controlled trials and meta-analysis. J Pineal Res. 2005 Nov;39(4):360-6. doi: 10.1111/j.1600-079X.2005.00258.x. PMID 16207291
- [Background] Seely D, Wu P, Fritz H, Kennedy DA, Tsui T, Seely AJ, Mills E. Melatonin as adjuvant cancer care with and without chemotherapy: a systematic review and meta-analysis of randomized trials. Integr Cancer Ther. 2012 Dec;11(4):293-303. doi: 10.1177/1534735411425484. Epub 2011 Oct 21. PMID 22019490
- [Derived] Seely D, Legacy M, Auer RC, Fazekas A, Delic E, Anstee C, Angka L, Kennedy MA, Tai LH, Zhang T, Maziak DE, Shamji FM, Sundaresan RS, Gilbert S, Villeneuve PJ, Ashrafi AS, Inculet R, Yasufuku K, Waddell TK, Finley C, Shargall Y, Plourde M, Fergusson DA, Ramsay T, Seely AJE. Adjuvant melatonin for the prevention of recurrence and mortality following lung cancer resection (AMPLCaRe): A randomized placebo controlled clinical trial. EClinicalMedicine. 2021 Feb 27;33:100763. doi: 10.1016/j.eclinm.2021.100763. eCollection 2021 Mar. PMID 33681747
- See also: The Canadian College of Naturopathic Medicine — http://www.ccnm.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: To receive 20 mg of melatonin nightly for 1 year
  melatonin: 20 mg ingested nightly
- Placebo: To receive matched supplement to the experimental arm in same schedule
  placebo: similar to experimental in all ways except for lack of active ingredient
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 356 | 353
Completed | 157 | 173
Not Completed | 199 | 180
Not completed — Cancer Recurrence | 58 | 58
Not completed — Withdrawal by Subject | 117 | 100
Not completed — Lost to Follow-up | 3 | 6
Not completed — Protocol Violation | 10 | 12
Not completed — Death | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Treatment: To receive 20 mg of melatonin nightly for 1 year
  melatonin: 20 mgs ingested nightly
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 356 | 353 | 709
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (8.5) | 67.2 (8.6) | 67.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 208 | 398
  Male | 166 | 145 | 311
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pre-Operative Chemotherapy or Radiation [Count of Participants; unit: Participants] | 8 | 14 | 22
Smoking History [Count of Participants; unit: Participants]
  Current Smoker | 47 | 52 | 99
  Past Smoker | 279 | 263 | 542
  Never Smoked | 25 | 31 | 56
  Unknown | 5 | 7 | 12
Histological Subtype [Count of Participants; unit: Participants]
  Squamous Cell | 93 | 72 | 165
  Adenocarcinoma | 229 | 239 | 468
  Large Cell | 7 | 15 | 22
  Bronchoalveolar | 10 | 8 | 18
  Undifferentiated | 2 | 3 | 5
  Other | 14 | 14 | 28
  Non-Surgical | 1 | 2 | 3
Incision Type [Count of Participants; unit: Participants]
  Minimally Invasive Surgery (MIS) | 213 | 212 | 425
  MIS Converted to Open | 27 | 19 | 46
  Open | 114 | 122 | 236
  Non-Surgical | 1 | 2 | 3
Surgery Type [Count of Participants; unit: Participants]
  Pneumonectomy | 16 | 21 | 37
  Lobectomy | 290 | 284 | 574
  Segmentectomy | 18 | 16 | 34
  Wedge Resection | 31 | 29 | 60
  No Operation | 1 | 3 | 4
Pathological Cancer Stage [Count of Participants; unit: Participants] — Overall 7th Edition American Joint Committee on Cancer (AJCC) stage (I-IV) based on the TNM classification. T refers to tumor size, N refers to nearby lymph nodes and M represents metastasized (spread) to other parts of the body. This staging number is obtained as a sum of the TNM classification. The lower the number, the lower the cancer stage and the better the prognosis for the patient. The higher the stage, the worse the prognosis.
  Participants
    Stage I | 245 | 217 | 462
    Stage II | 75 | 92 | 167
    Stage III | 32 | 38 | 70
    Stage IV | 2 | 3 | 5
    Non-Surgical | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Lung Cancer Recurrence or Mortality - 2 Years
Description: Disease-Free survival (DFS) at 2 years post-surgery. DFS is measured by the number of participants in both arms who have experienced a recurrence OR mortality at 2 years.
Time Frame: 2 years
Population: Intention to treat - all participants analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Melatonin: To receive 20 mg of melatonin nightly for 1 year following surgery.
- Placebo: To receive 20 mg placebo nightly for 1 year following surgery
  placebo: similar to experimental in all ways except for lack of active ingredient
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 356 | 353
Participants | 80 | 85
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Analysis conducted was an adjusted logistic regression (adjuvant chemotherapy, adjuvant radiation, smoking history). Results were presented as a relative risk. Based on an estimated 30% outcome rate of recurrence or mortality in the control arm, 294 participants per arm provided 80% power to detect a relative risk of one third at an alpha of 0.05. We inflated this sample size to 346 per arm to account for 15% lost to follow-up; Test type: Superiority; p = 0.94, Regression, Logistic; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.83 to 1.22]

2. Secondary Outcome: Quality of Life
Description: Participant-reported quality of life using the European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire C-30 (EORTC QLQ C-30) and Lung Cancer 13 (EORTC QLQ LC13) questionnaires. Scores represent a value from 0-100. Symptom and LC13 scale: 0 represents best health, 100 worst health. Global and functional scales: 100 represents best health, 0 represents worst health. Full scoring algorithms available here: https://www.eortc.org/app/uploads/sites/2/2018/02/SCmanual.pdf
Time Frame: 2 years
Population: Intention to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale of 0-100
Groups:
- Melatonin: To receive 20 mg of melatonin nightly for 1 year post surgery
- Placebo: To receive 20 mg placebo nightly for 1 year post surgery
  placebo: similar to experimental in all ways except for lack of active ingredient
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 356 | 353
Score on a scale of 0-100
  Symptom Scale (Baseline) | 21.4 [19.1 to 23.7] | 20.3 [18.0 to 22.6]
  Symptom Scale (1Y) | 18.2 [15.7 to 20.7] | 17.0 [14.3 to 19.5]
  Symptom Scale (2Y) | 17.3 [14.6 to 20.0] | 15.8 [13.2 to 18.5]
  Functional Scale (Baseline) | 75.8 [73.2 to 78.5] | 75.5 [72.9 to 78.2]
  Functional Scale (1Y) | 79.9 [77.0 to 82.8] | 81.1 [78.2 to 84.1]
  Functional Scale (2Y) | 80.2 [77.0 to 83.3] | 80.5 [77.4 to 83.7]
  Global Scale (Baseline) | 64.5 [61.3 to 67.8] | 62.7 [59.5 to 66.0]
  Global Scale (1Y) | 69.6 [65.9 to 73.3] | 71.6 [67.9 to 75.3]
  Global Scale (2Y) | 70.7 [66.7 to 74.7] | 72.7 [68.8 to 76.7]
  LC13 Scale (Baseline) | 17.4 [15.3 to 19.4] | 19.0 [17.0 to 21.0]
  LC13 Scale (1Y) | 17.8 [15.5 to 20.0] | 18.1 [15.9 to 20.4]
  LC13 Scale (2Y) | 17.1 [14.7 to 19.5] | 17.5 [15.2 to 19.9]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Analysis for the LC-13 scale; Test type: Superiority; p = 0.36, Mixed Models Analysis; Between-arm least squares mean difference in change from randomization to 24 months post-surgery represented the effect of the intervention; Mean Difference (Net) = 1.2, 95% CI 2-sided [-1.3 to 3.7]
Statistical Analysis 2: Comparison: Melatonin vs Placebo; Analysis for Symptom Scale; Test type: Superiority; p = 0.80, Mixed Models Analysis — Between-arm least squares mean difference in change from randomization to 24 months post-surgery represented the effect of the intervention; Mean Difference (Net) = 0.4, 95% CI 2-sided [-2.5 to 3.3]
Statistical Analysis 3: Comparison: Melatonin vs Placebo; Analysis for Functional Scale; Test type: Superiority; p = 0.69, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Net) = -0.7, 95% CI 2-sided [-4.1 to 2.7]
Statistical Analysis 4: Comparison: Melatonin vs Placebo; Analysis for Global Scale; Test type: Superiority; p = 0.11, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Net) = -3.8, 95% CI 2-sided [-8.5 to 0.9]

3. Secondary Outcome: Fatigue
Description: Measured using the Multidimensional Fatigue Inventory 20 (MFI-20) questionnaire. Scores are on a scale of 0-100, where 100 is the best health and 0 is the worst health.
Time Frame: 2 years
Population: Intention to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale of 0-100
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 356 | 353
Score on a scale of 0-100
  Baseline | 59.8 [56.3 to 62.9] | 57.0 [53.8 to 60.1]
  1Y | 61.4 [57.9 to 64.9] | 62.4 [58.9 to 65.9]
  2Y | 62.7 [59.0 to 66.5] | 63.1 [59.4 to 66.8]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Between-arm least squares mean difference in change from randomization to 24 months post-surgery represented the effect of the intervention; Test type: Superiority; p = 0.13, Mixed Models Analysis; Mean Difference (Net) = -3.1, 95% CI 2-sided [-7.2 to 0.9]

4. Secondary Outcome: Sleep
Description: Measured using the Medical Outcomes Study (MOS) Sleep Survey. Scales used were Sleep Adequacy and Sleep problems Index II. Scores are on a scale of 0-100. Sleep Adequacy: 100 represents best health; 0 represents worst health. Problems index: 0 represents best health; 100 represents worst health.
Time Frame: 2 years
Population: Intention to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale of 0-100
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 356 | 353
Score on a scale of 0-100
  Sleep Adequacy (Baseline) | 56.7 [52.5 to 61.0] | 53.8 [49.5 to 58.0]
  Sleep Adequacy (1Y) | 60.9 [56.1 to 65.7] | 61.5 [56.7 to 66.3]
  Sleep Adequacy (2Y) | 59.4 [54.2 to 64.5] | 60.5 [55.4 to 65.5]
  Sleep Problems Index II (baseline) | 32.7 [29.9 to 35.6] | 33.6 [30.8 to 36.4]
  Sleep Problems Index II (1Y) | 28.0 [24.9 to 31.2] | 27.7 [24.5 to 30.8]
  Sleep Problems Index II (2Y) | 27.5 [24.2 to 30.8] | 26.9 [23.6 to 30.2]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Sleep Adequacy Analysis; Test type: Superiority; p = 0.18, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -4.1, 95% CI 2-sided [-10.0 to 1.9]
Statistical Analysis 2: Comparison: Melatonin vs Placebo; Sleep problems index II analysis; Test type: Superiority; p = 0.41, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 1.4, 95% CI 2-sided [-2.0 to 4.8]

5. Secondary Outcome: Pain Levels
Description: Calculated using the Brief Pain Inventory. Each scale ranges from 0-10, where 0 is no pain and 10 is the worst possible pain.
Time Frame: 3 months
Population: Only those recruited from the Ottawa Hospital were included in this analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale of 0-10
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 156 | 157
Score on a scale of 0-10
  Baseline | 2.4 (2.4) | 2.3 (2.2)
  3 months | 2.3 (2.1) | 2.4 (2.2)

6. Secondary Outcome: Anxiety
Description: Measured using the Beck Anxiety Inventory. Scored range from 0-63, where 0 is no anxiety and 63 is the worst possible anxiety.
Time Frame: 2 years
Population: Only participants recruited from The Ottawa Hospital were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale of 0-63
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 156 | 157
Score on a scale of 0-63
  Baseline | 8.2 (8.5) | 8.3 (8.4)
  2Y | 6.2 (6.9) | 6.4 (7.6)

7. Secondary Outcome: Depression
Description: Measured using the Beck Depression Inventory II. Scores range from 0-63, where 0 is no depression and 63 is the worst possible depression.
Time Frame: 2 years
Population: Only participants recruited from The Ottawa Hospital were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale of 0-63
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 156 | 157
Score on a scale of 0-63
  Baseline | 8.1 (7.2) | 8.6 (8.5)
  2Y | 6.6 (5.9) | 7.7 (8.0)

8. Secondary Outcome: Adverse Events (Chemotherapy)
Description: Number of participants who experienced an adverse event related to their adjuvant chemotherapy
Time Frame: 2 years
Population: Only those who received adjuvant chemotherapy were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 66 | 68
Participants | 44 | 48
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority; p = 0.62, Chi-squared

9. Secondary Outcome: Lung Cancer Recurrence or Mortality - 5 Years
Description: Measured as disease-free survival (DFS) at 5 years. DFS was measured by the incidence of a recurrence OR mortality up to 5 years post-surgery.
Time Frame: up to 5 years
Population: Intention to treat - all participants analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 356 | 353
Participants
  All participants | 133 | 130
  Early Stage Cancer: number analyzed (Participants) | 320 | 309
  Early Stage Cancer | 109 | 99
  Late Stage Cancer: number analyzed (Participants) | 34 | 41
  Late Stage Cancer | 23 | 31
Statistical Analysis 1: Comparison: Melatonin vs Placebo; DFS up to five years post-surgery was compared using Kaplan-Meier curves and the log rank test, followed by a hazard ratio calculated using the Cox proportional hazard model adjusting for adjuvant chemotherapy, adjuvant radiation, and smoking history; Test type: Superiority; p = 0.41, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.85 to 1.07]
Statistical Analysis 2: Comparison: Melatonin vs Placebo; This analysis included only those with stage I or II cancer (pathologic stage). DFS up to five years post-surgery was compared using Kaplan-Meier curves and the log rank test, followed by a hazard ratio calculated using the Cox proportional hazard model adjusting for adjuvant chemotherapy, adjuvant radiation, and smoking history; Test type: Superiority; p = 0.66, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.85 to 1.11]
Statistical Analysis 3: Comparison: Melatonin vs Placebo; This analysis included only those participants who had stage III or IV cancer (pathologic stage). DFS up to five years post-surgery was compared using Kaplan-Meier curves and the log rank test, followed by a hazard ratio calculated using the Cox proportional hazard model adjusting for adjuvant chemotherapy, adjuvant radiation, and smoking history; Test type: Superiority; p = 0.004, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.61 to 0.92]

10. Secondary Outcome: Blood Tests to Examine the Effects of Melatonin on the Immune System (Raw Values)
Description: NK cell cytotoxicity changes from baseline to 6 months
Time Frame: 6 months
Population: Participants who qualified for the sub-study only.
Measure: Mean (Standard Error); unit: Percent killing of K62 cells
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 35 | 37
Percent killing of K62 cells
  Cytotoxicity (baseline) | 49.8 (3.6) | 42.7 (3.3)
  Cytotoxicity (6 months) | 49.2 (3.0) | 46.4 (3.8)
Statistical Analysis 1: Comparison: Melatonin; Analysis of melatonin changes; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-3.21 to 4.56]
Statistical Analysis 2: Comparison: Placebo; Analysis of placebo changes; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3.63, 95% CI 2-sided [-0.15 to 7.42]

11. Secondary Outcome: Adverse Events (Radiation)
Description: Number of participants who experienced an adverse event related to their adjuvant radiation therapy
Time Frame: 2 years
Population: Only those who received adjuvant radiation were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 22 | 21
Participants | 8 | 5
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority; p = 0.37, Chi-squared

12. Secondary Outcome: Blood Tests to Examine the Effects of Melatonin on the Immune System (Comparison Between Groups)
Description: Differences in NK cell cytotoxicity between both arms
Time Frame: 6 months
Population: Only those who were enrolled in the sub study and qualified for analysis were included.
Measure: Mean (95% Confidence Interval); unit: Ratio of percent cytotoxicity
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 35 | 37
Ratio of percent cytotoxicity | 1.1 [0.97 to 1.23] | 1.16 [0.96 to 1.37]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; This analysis compares the mean ratios of 6 month cytotoxicity and baseline cytotoxicity between arms; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 2 Years
Description: An adverse event is any untoward medical occurrence in a patient administered a medicinal product which does not necessarily have to have a causal relationship with this treatment. A serious adverse event is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or results in prolonging of existing hospitalization, results in a persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Arm/Group | Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 95/356 | 91/353
Serious Adverse Events (participants affected / at risk) | 84/356 | 89/353
Other Adverse Events (participants affected / at risk) | 184/356 | 166/353
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melatonin (N=356) | Placebo (N=353)
Hypercalcemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Angina (Cardiac disorders) | 0 | 1
Aortic Valve Replacement (Cardiac disorders) | 1 | 0
Apical thrombosis (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
NSTEMI (Cardiac disorders) | 0 | 2
Pericardial Effusion (Cardiac disorders) | 1 | 0
STEMI (Cardiac disorders) | 1 | 0
Left para-opthalmic aneurysm (Eye disorders) | 0 | 1
Retinal Tear (Eye disorders) | 1 | 0
Adbominal Abcess (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gall bladder removal (Gastrointestinal disorders) | 1 | 1
Lower GI Bleeding (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Perforated Bowel (Gastrointestinal disorders) | 1 | 0
SBO (Gastrointestinal disorders) | 0 | 1
Upper GI bleeding (Gastrointestinal disorders) | 1 | 0
Dehydration (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Chest Infection (Infections and infestations) | 1 | 0
Fever (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Injury, poisoning and procedural complications) | 1 | 1
Back sprain (Injury, poisoning and procedural complications) | 1 | 0
Broken elbow (Injury, poisoning and procedural complications) | 0 | 1
Discitis (Injury, poisoning and procedural complications) | 1 | 0
Hip replacement surgery (Injury, poisoning and procedural complications) | 2 | 0
Left above-knee amputation (Injury, poisoning and procedural complications) | 1 | 0
Left total knee arthroplasty (Injury, poisoning and procedural complications) | 1 | 0
Osteophyte fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella and fibular fracture (Injury, poisoning and procedural complications) | 1 | 0
Shoulder Replacement Surgery (Injury, poisoning and procedural complications) | 1 | 0
Toe Amputation (Injury, poisoning and procedural complications) | 0 | 1
Weakness (Injury, poisoning and procedural complications) | 1 | 0
Bladder Cancer Recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
New Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
New Neoplasm - Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
New Neoplasm - Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
New Neoplasm - Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
New Neoplasm - Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
New Neoplasm - Medullary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
New Neoplasm - Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
New Neoplasm - Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
New Neoplasm - Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
New Neoplasm - thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
New Neoplasm - thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
New Neoplasm - Urothelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pericarditis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Leptomeningeal disease (Nervous system disorders) | 1 | 0
Neuro-syncope (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0
Acute renal failure (Renal and urinary disorders) | 1 | 0
Diabetic ketoacidosis (Renal and urinary disorders) | 1 | 0
Renal Caliculi (Renal and urinary disorders) | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 1 | 1
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death (Respiratory, thoracic and mediastinal disorders) | 37 | 37
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Empyema (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Prolonged Air Leak (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subcutaneous Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Aneurism Surgery (Surgical and medical procedures) | 0 | 1
Completion thyroidectomy (Surgical and medical procedures) | 0 | 1
Resection of Liposarcoma (Surgical and medical procedures) | 1 | 0
Thoracotomy (Surgical and medical procedures) | 0 | 1
Total thyroidectomy (Surgical and medical procedures) | 0 | 1
Peripheral Ischemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melatonin (N=356) | Placebo (N=353)
Anemia (Blood and lymphatic system disorders) | 2 | 3
Blood/bone marrow - Other (myelotoxicity) (Blood and lymphatic system disorders) | 0 | 1
Elevated ALT (Blood and lymphatic system disorders) | 0 | 1
ELevated AST (Blood and lymphatic system disorders) | 0 | 1
Elevated creatinine levels (Blood and lymphatic system disorders) | 1 | 0
Elevated TNI (Blood and lymphatic system disorders) | 0 | 1
Hyperglycemia (Blood and lymphatic system disorders) | 2 | 1
Hypokalemia (Blood and lymphatic system disorders) | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 12 | 7
Thrombic event (Blood and lymphatic system disorders) | 0 | 1
Angina (Cardiac disorders) | 0 | 2
Atrial Arrhythmia (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 1
Cardiac - Intra-Op Bleeding (Cardiac disorders) | 1 | 0
Cardiac Embolism (Cardiac disorders) | 0 | 1
Coronary Artery Calcification (Cardiac disorders) | 1 | 0
Heart Palpitations (Cardiac disorders) | 1 | 1
Hypertension (Cardiac disorders) | 2 | 0
Hypotension (Cardiac disorders) | 1 | 2
Syncope (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 5 | 0
Thoracic Aortic Calcification (Cardiac disorders) | 1 | 0
Hearing loss (Ear and labyrinth disorders) | 3 | 1
Hot swollen ears (Ear and labyrinth disorders) | 0 | 1
ruptured eardrum (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 7
Hyperthyroidism (Endocrine disorders) | 1 | 0
Blurred Vision (Eye disorders) | 1 | 1
Burning eyes (Eye disorders) | 1 | 0
Cataracts (Eye disorders) | 1 | 0
decreased vision in left eye (Eye disorders) | 0 | 1
Itchiness of eyes (Eye disorders) | 1 | 0
Left eye pain (after starting chemo) (Eye disorders) | 0 | 1
Vision changes (Eye disorders) | 1 | 0
Vitreous detachment/flashing lights (Eye disorders) | 1 | 0
Abdominal bloating (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 6
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Acid reflux (Gastrointestinal disorders) | 2 | 1
Appetite changes (Gastrointestinal disorders) | 6 | 8
Bloating (Gastrointestinal disorders) | 1 | 3
Burping (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 16 | 16
Diarrhea (Gastrointestinal disorders) | 29 | 18
Dilaudid related withdrawal symptoms (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 2
Esophagitis (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 3 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
GERD (Gastrointestinal disorders) | 3 | 3
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileostomy reversal (Gastrointestinal disorders) | 0 | 1
Indigestion (Gastrointestinal disorders) | 4 | 0
Mouth Ulcers (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 31 | 34
Odynophagia (Gastrointestinal disorders) | 0 | 1
Thrush (mouth) (Gastrointestinal disorders) | 2 | 0
UGI Bleeding (Gastrointestinal disorders) | 0 | 1
Ulcerative colitis flare up (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 11 | 8
Allergic Reaction (General disorders) | 1 | 2
Costovertebral angle tenderness (General disorders) | 0 | 1
Dehydration (General disorders) | 1 | 1
Desaturation (General disorders) | 0 | 2
Failure to thrive (General disorders) | 0 | 1
Fatgiue (General disorders) | 56 | 56
Generally unwell (General disorders) | 0 | 1
Hair loss (General disorders) | 1 | 0
Hot flashes (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Left vocal cord swelling (General disorders) | 0 | 1
Loss of voice (General disorders) | 0 | 2
Night sweats (General disorders) | 1 | 1
Peripheral Edema (General disorders) | 4 | 2
Phlebitis (General disorders) | 1 | 0
Restlessness (General disorders) | 0 | 1
Ulcer on tongue (General disorders) | 1 | 0
Voice hoarseness (General disorders) | 1 | 3
Weakness (General disorders) | 1 | 0
Weight gain (General disorders) | 1 | 3
Weight loss (General disorders) | 2 | 2
Gall bladder attack (Hepatobiliary disorders) | 2 | 0
bladder infection (Infections and infestations) | 1 | 1
C-Difficile (Infections and infestations) | 2 | 0
Chest infection (Infections and infestations) | 1 | 1
Cold/Flu Symptoms (Infections and infestations) | 7 | 13
Fever (Infections and infestations) | 1 | 0
Fungal lung infection (Aspergillus) (Infections and infestations) | 0 | 1
Infectious Sebaceous Cyst (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Oral candida infection (Infections and infestations) | 0 | 1
pelvic sepsis (Infections and infestations) | 1 | 0
Shingles (Infections and infestations) | 1 | 0
Sinus infection (Infections and infestations) | 3 | 0
skin infection (Infections and infestations) | 0 | 4
Surgical site infection (Infections and infestations) | 2 | 0
Throat Infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Back of tongue pain (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Injury, poisoning and procedural complications) | 2 | 6
Bone pain in upper thigh (Injury, poisoning and procedural complications) | 0 | 1
Burn marks (arm) (Injury, poisoning and procedural complications) | 0 | 1
Burning sensation of feet, mostly at night (Injury, poisoning and procedural complications) | 0 | 1
Burning sensation when going to bathroom (Injury, poisoning and procedural complications) | 0 | 1
Calf pain at night after starting chemo (Injury, poisoning and procedural complications) | 1 | 0
Chronic pain/post-thoracotomy discomfort (Injury, poisoning and procedural complications) | 0 | 1
elbow pain (left) (Injury, poisoning and procedural complications) | 0 | 1
Erythema and tenderness arm, site of IV needle (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2
Fracture - nose (Injury, poisoning and procedural complications) | 0 | 1
Fracture - wrist (Injury, poisoning and procedural complications) | 0 | 1
Fractured foot (Injury, poisoning and procedural complications) | 0 | 1
Fractures (Injury, poisoning and procedural complications) | 0 | 1
Joint pain (Injury, poisoning and procedural complications) | 0 | 1
Laceration - left fingers (Injury, poisoning and procedural complications) | 0 | 1
Left arm pain while on chemo (Injury, poisoning and procedural complications) | 0 | 1
Left hand tingling (Injury, poisoning and procedural complications) | 1 | 0
Left leg numbness (Injury, poisoning and procedural complications) | 1 | 0
Left shoulder and neck pain (Injury, poisoning and procedural complications) | 1 | 0
leg cramps (Injury, poisoning and procedural complications) | 1 | 0
Leg/joint pain (Injury, poisoning and procedural complications) | 1 | 0
Lower back pain (Injury, poisoning and procedural complications) | 0 | 1
Pain (Injury, poisoning and procedural complications) | 5 | 5
Pain (back) (Injury, poisoning and procedural complications) | 1 | 0
Pain (leg) (Injury, poisoning and procedural complications) | 0 | 1
Pain (ongoing issue from fibromyalgia) (Injury, poisoning and procedural complications) | 0 | 1
Pain in left foot (Injury, poisoning and procedural complications) | 1 | 0
Pain in right side (tender to touch) (Injury, poisoning and procedural complications) | 1 | 0
Pain in right side flank (Injury, poisoning and procedural complications) | 0 | 1
pain left leg (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Pain (Injury, poisoning and procedural complications) | 18 | 16
R. Arm weakness (Injury, poisoning and procedural complications) | 1 | 0
Right arm weakness (Injury, poisoning and procedural complications) | 1 | 0
Severe stabbing pain in thighs (Injury, poisoning and procedural complications) | 0 | 1
Shoulder pain (Injury, poisoning and procedural complications) | 1 | 2
Sore back (Injury, poisoning and procedural complications) | 0 | 1
Sprained ankle (Injury, poisoning and procedural complications) | 1 | 0
Surgical Site Pain (Injury, poisoning and procedural complications) | 2 | 7
Swollen right hand (pain Rt 2 fingers) (Injury, poisoning and procedural complications) | 1 | 0
Tenderness to incision site (Injury, poisoning and procedural complications) | 1 | 0
Tooth Infection (Injury, poisoning and procedural complications) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
inflammatory pseudo tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
New Neoplasm - breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
New Neoplasm - Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
New Neoplasm - Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
New Neoplasm - pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
New Neoplasm - Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
New Neoplasm - Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cognitive dysfunction/loss of memory (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 7 | 5
Drowsiness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 11 | 14
Hyperarousal (Nervous system disorders) | 1 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Lighheadedness (Nervous system disorders) | 1 | 1
loss of balance (Nervous system disorders) | 0 | 1
Memory difficulty (Nervous system disorders) | 1 | 0
Migrane (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 2
Peripheral Neuropathy (Nervous system disorders) | 9 | 3
Restlessness leg syndrome (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Sensory neuropathy (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 3
Spacey feeling (Nervous system disorders) | 0 | 1
Spinal Stenosis (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Subcostal neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 4 | 1
Vertigo (Nervous system disorders) | 3 | 2
Vivid Dreams (Nervous system disorders) | 0 | 3
Anorexia (Psychiatric disorders) | 3 | 7
Anxiety (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 4 | 5
Hallucinations (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 39 | 36
Anal fissures (Renal and urinary disorders) | 0 | 1
burning sensation when urinating (Renal and urinary disorders) | 1 | 0
Difficulty Urinating (Renal and urinary disorders) | 1 | 1
Frequent urination (Renal and urinary disorders) | 1 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
L. Kidney Cyst (Renal and urinary disorders) | 1 | 0
Discomfort or pain - breast area Rt side (Reproductive system and breast disorders) | 0 | 1
Pain - right breast (dense feeling) (Reproductive system and breast disorders) | 1 | 0
Prolapsed uterus (Reproductive system and breast disorders) | 0 | 1
Ulceration vagina mucosa (Reproductive system and breast disorders) | 1 | 0
Air Leak (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Bonchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Burning sensation back of throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 6 | 9
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 33 | 19
Empyema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Fungal lung infection (Aspergillus) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiatal Hernia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease progression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Mucus in chest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Radiation pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rib fractures (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Separated rib (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Subcutaneous Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
dry mouth (Skin and subcutaneous tissue disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Increased thickness in nails (Skin and subcutaneous tissue disorders) | 1 | 0
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 | 0
Left vocal cord swelling (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 16
Sclera derma (Skin and subcutaneous tissue disorders) | 1 | 0
skin eruptions (Skin and subcutaneous tissue disorders) | 0 | 1
Gall bladder removal (Surgical and medical procedures) | 1 | 0
Hernia (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT00668707/Prot_SAP_000.pdf